CLINICAL TRIAL: NCT02228109
Title: Multifocal Lens Centration and Its Effect on Visual Performance in a Presbyopic Population
Acronym: BUICK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Collaborators: Johnson & Johnson Vision Care (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 20067
Record Dates: First submitted 2014-08-26; First posted 2014-08-28 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Acuvue Oasys for Presbyopia (Experimental): Acuvue Oasys for Presbyopia contact lenses worn
  Interventions: Device: Acuvue Oasys for Presbyopia
- PureVision2 for Presbyopia (Experimental): PureVision2 for Presbyopia contact lenses worn
  Interventions: Device: PureVision2 for Presbyopia
- Biofinity Multifocal (Experimental): Biofinity Multifocal contact lenses worn
  Interventions: Device: Biofinity Multifocal

INTERVENTIONS:
Device: Acuvue Oasys for Presbyopia — Acuvue Oasys for Presbyopia contact lenses worn
  Arms: Acuvue Oasys for Presbyopia
Device: PureVision2 for Presbyopia — PureVision2 for Presbyopia contact lenses worn
  Arms: PureVision2 for Presbyopia
Device: Biofinity Multifocal — Biofinity Multifocal contact lenses worn
  Arms: Biofinity Multifocal

SUMMARY:
The purpose of this study is to use a corneal topographer, a device that is readily available in most optometric practices, in order to determine the position of the multifocal (MF) contact lens (CL) optics in relation to the optics of the eye. The specific purpose of this study is to evaluate if there is a relationship between the positioning of the optics of the study lenses and the objective and subjective visual performance as well as participant satisfaction. The MF CL lenses will be fitted to two groups of participants (previously unsuccessful vs. currently successful MF CL wearers).

HYPOTHESES

* The measurement of the power distribution acquired from the Medmont E300 corneal topographer is effective in determining MF CL lens centration and is a predictor of MF CL success.
* There is a difference in MF CL centration, determined by corneal topography, between successful and unsuccessful MF CL wearers.
* MF CL centration, determined by corneal topography, is correlated with visual performance, determined by ocular aberrometry, measures of visual acuity and subjective satisfaction.

ELIGIBILITY:
Inclusion Criteria:

A person is eligible for inclusion in the study if he/she:

1. Is at least 42 years of age and has full legal capacity to volunteer;
2. Has read and signed an information consent letter;
3. Is willing and able to follow instructions and maintain the appointment schedule;
4. Has previous experience with wearing MF CLs;
5. Is able to be successfully fitted with all study lenses;
6. Has a vertex-corrected spherical distance prescription of +6.00 to 8.00D (inclusive) in both eyes;
7. Has a spectacle cylinder ≤0.75D in both eyes;
8. Requires a reading addition of ≥+1.00D;

Exclusion Criteria:

A person will be excluded from the study if he/she:

1. Is participating in any concurrent clinical or research study;
2. Has any known active* ocular disease and/or infection;
3. Has a systemic condition that in the opinion of the investigator may affect a study outcome variable;
4. Is using any systemic or topical medications that in the opinion of the investigator may affect a study outcome variable;
5. Has a known sensitivity to the diagnostic pharmaceuticals to be used in the study;
6. Is pregnant, lactating or planning a pregnancy at the time of enrolment;
7. Is aphakic;
8. Has undergone refractive error surgery;
9. Has monocular best-corrected VA of worse than 20/30 in each eye;
10. Has amblyopia or strabismus;
11. Has anisometropia >2D between both eyes

    * For the purposes of this study, active ocular disease is defined as infection or inflammation which requires therapeutic treatment. Mild (i.e. not considered clinically relevant) lid abnormalities (blepharitis, meibomian gland dysfunction, papillae), corneal and conjunctival staining and dry eye are not considered active ocular disease. Neovascularization and corneal scars are the result of previous hypoxia, infection or inflammation and are therefore not active.

Min Age: 42 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-12; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Decentration | Day 1
  Decentration (in mm and axis of decentration) of the multifocal contact lens optical center relative to ocular reference points (e.g. the pupil center or the line of sight), determined using difference maps produced by the Medmont E300 corneal topographer.

SECONDARY OUTCOMES:
Visual Acuity (high contrast) at distance | Day 1
  Visual Acuity (high contrast) (logMAR) at distance 6m
Visual Acuity (high contrast) at intermediate distance | Day 1
  Visual Acuity (high contrast) (logMAR) at intermediate distance 1m
Visual Acuity (high contrast) at near | Day 1
  Visual Acuity (high contrast) (logMAR) at near (0.4m)
Visual Acuity (low contrast) at distance | Day 1
  Visual Acuity (low contrast) at distance 6m
Visual Acuity (low contrast) at intermediate distance | Day 1
  Visual Acuity (low contrast) (logMAR) at intermediate distance 1m
Visual Acuity (low contrast) at near | Day 1
  Visual Acuity (low contrast) (logMAR) at near (0.4m)
Overall subjective rating of lens performance in real world tasks | Day 1
  Participants rate overall satisfaction with vision with the contact lenses on a scale of 0-100, where 0=completely dissatisfied and 100=completely satisfied, after completing a series of real world tasks.
Ocular aberrometry | Day 1
  Ocular aberrometry as measured by a LADARWave aberrometer

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, PhD, Principal Investigator — CCLR, University of Waterloo
Locations (1):
- Centre for Contact Lens Research, University of Waterloo, Waterloo, Ontario, Canada